CLINICAL TRIAL: NCT06086301
Title: Pilot Testing Post-Intensive Care Transitions Using Rehabilitation and Engagement To Heal ICU Survivors and Families (PICTURE-THIS)
Brief Title: Pilot Testing PICTURE-THIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Leslie Scheunemann, Assistant Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY23010154; K08HS027210 (AHRQ)
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Post-intensive Care Syndrome; Transitional Care; Critical Care; Health Services
Keywords: Pilot Study; Critical Illness Survivors; Family Caregivers; Transitional care; Rehabilitation; Family Support
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICTURE-THIS services (Experimental): This group receives a Run-In Phase followed by outpatient transitional care management (up to 8 visits over 3 months), activity-based rehabilitation (up to 10 visits over 3 months), and social support for patients and families (ongoing screening and referral). They will also undergo outcome assessments at discharge, 3 and 6 months.
  Interventions: Other: PICTURE-THIS; Behavioral: Run-In Phase
- Enhanced Usual Care (Active Comparator): Enhanced Usual Care (EUC) control group will rececive a Run-in Phase followed by an informational brochure with regular assessments on the same schedule as the PICTURE-THIS group (i.e., discharge, 3 and 6 months)
  Interventions: Other: Enhanced Usual Care; Behavioral: Run-In Phase

INTERVENTIONS:
Other: PICTURE-THIS — Discharge plans include scheduling post-discharge appointments, community support referrals, transportation arrangements, and addressing identified gaps. Transition care includes 8 check-ins over 3 months post-discharge, focusing on assessing, troubleshooting, and celebrating transition successes, using phone or video. Telehealth-assisted 'warm hand-offs' will connect interventionists with home health and primary care teams during initial visits. '1st touch daytime troubleshooting' offers extra support between check-ins. Problem-solving rehabilitation will be continued from hospital to home, with 7-10 sessions over 3 months, including a home safety survey. A Post-ICU Caregiver Toolkit provides workbooks, training videos, and resources. Lastly, referrals for patient and caregiver social/mental health support are provided.
  Arms: PICTURE-THIS services
Other: Enhanced Usual Care — Enhanced Usual Care (EUC) control group will receive: (1) Patient and Family Re-sources published by the SCCM for PICS prior to hospital discharge; (2) ongoing assessments on the same schedule as the PICTURE-THIS intervention; (3) referral for urgent or emergent issues identified during assessments. The investigators will not provide the URL for the Post-ICU Caregiving Toolkit but the investigators will not restrict its access either. This control design balances 3 goals: 1) masking participants to group allocation; 2) responding ethically to harm/distress; 3) maintaining group separation to optimize efficacy testing of PICTURE-THIS.
  Arms: Enhanced Usual Care
Behavioral: Run-In Phase — All participants receive a Run-In Phase during the acute critical illness hospitalization. It consists of 3 inpatient study visits: (1) health and social screening; (2) planning for rehabilitation; (3) discharge education and training.

SUMMARY:
This is a single-center pilot study examining the feasibility and acceptability of a transitional rehabilitation intervention, PICTURE-THIS, among critical illness survivors and their families. The intervention activities include transitional care coordination and activity-based rehabilitation delivered by a specialist team and integrated into usual care. There are three components to the assessment of feasibility and acceptability in this study:

1. User testing the PICTURE-THIS protocol to work out basic challenges to feasibility and acceptability.
2. Assessing the feasibility and acceptability of the user-tested PICTURE-THIS protocol.
3. Assessing the feasibility and acceptability of research activities required to test the clinical efficacy of PICTURE-THIS to improve outcomes among critical illness survivors and their family caregivers.

DETAILED DESCRIPTION:
Purpose: PICTURE-THIS is a transitional rehabilitation intervention for critical illness survivors and their family caregivers. It has 2 phases: (1) A Run-In Phase in the hospital; (2) A post-discharge phase. The purpose of this study is to user- and pilot-test the protocols for PICTURE-THIS.

Aim 1: To test, troubleshoot, and revise study procedures and protocols for PICTURE-THIS with a convenience sample of critical illness survivors and their family caregivers.

The investigators will: 1) ensure that dyads reliably adhere to PICTURE-THIS protocols; 2) troubleshoot assessments at enrollment and 3 and 6 month follow-up; 3) refine data collection and management procedures.

Aim 2: To pilot test PICTURE-THIS for feasibility and acceptability among a convenience sample of critical illness survivors and their family caregivers.

Feasibility will be demonstrated by: 1) >80% completion of clinical assessments; 2) >80% retention rate (enrolled patients attending ≥ 2 outpatient transitional care visits and 8 rehabilitation sessions); 2) >80% completion rate for surveys assessing outcomes.

Acceptability will be demonstrated by: 1) >80% participants being willing to recommend PICTURE-THIS to others; 2) >80% global acceptability survey score.

Feasibility and acceptability will be similar in participants living in rural communities compared to those living in urban/suburban ones.

Over half of critical illness survivors develop the Post-Intensive Care Syndrome (PICS), including long-lasting physical, cognitive, and psychological impairments. Without universal transitional care infrastructure, survivors and their families have high rates of unmet needs that result in: (1) adverse events including falls, caregiver stress, rehospitalizations, death and associated with high utilization of healthcare resources; (2) poor long-term outcomes including high symptom burden and reduced quality of life; (3) health disparities related to age, disability status, and income.

Addressing their transitional care needs in the post-ICU context requires a pragmatic, accessible, scalable intervention model. While Critical Illness Recovery Clinics are important hubs of innovation in PICS care, they are not accessible or scalable to meet the public health need which includes >3 million people in the United States each year. Further, they have not taken advantage of the rich intervention models from the field of transitional care to address care coordination and social needs early after critical illness. Our preliminary research showed that these intervention models can and should be adapted to the post-ICU context. It also suggested that adaptations should incorporate strengths-based rehabilitation interventions aimed at generating a virtuous cycle between mechanisms (e.g., mastery) and outcomes (e.g., participation in meaningful activities) to achieve multidomain wellbeing. Finally, the investigators and others showed that social determinants of health are ubiquitous factors in post-ICU care delivery that must be incorporated into intervention design.

To meet these needs, the investigators adapted evidence-based transitional care, activity-based rehabilitation, and family caregiving interventions into a single intervention called Post-Intensive Care Transitions Using Rehabilitation and Engagement To Heal ICU Survivors and Families (PICTURE-THIS). PICTURE-THIS is delivered by an interdisciplinary team that nimbly supports medical, nursing, rehabilitation, and social care needs in collaboration with existing hospital, home health, and primary care infrastructure. The purpose of this research study is to user and pilot test PICTURE-THIS prior to efficacy testing.

ELIGIBILITY:
Inclusion Criteria for Patient Participants:

≥50 years old. Admitted from home. Spend ≥48 hours in an ICU. Have an attending prognosis ≥ 12 months. Have some risk of ongoing functional impairment, indicated by a recorded HLM (Highest Level Mobility) < 8, AMPAC (Activity Measures for Post-Acute Care) < 24, or ICDSC (Intensive Care Delirium Screening Checklist) >2.

Exclusion Criteria for Patient Participants:

No identified caregiver. Unable to participate in English. Resides outside of Pennsylvania.

Inclusion Criteria for Family caregiver Participants:

≥21 years old. English-speaking. Providing support to the patient since the ICU stay

Exclusion Criteria for Family Caregiver Participants:

None

Inclusion Criteria for Healthcare Provider Participants:

Providing health services to a PICTURE-THIS dyad Willing to complete a survey

Exclusion Criteria for Healthcare Provider Participants:

None

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Enrollment | Up to 6 months
  Achieving an enrollment rate of 80% of eligible participants.
  Enrollment Rate (%) = (Number of Enrolled Participants / Number of Eligible Participants) x 100
Retention | Up to 6 months
  Maintaining an active engagement and complete participation rate of 80% throughout the study.
  Retention Rate (%) = (Number of Retained Participants / Number of Enrolled Participants) x 100

SECONDARY OUTCOMES:
PROPr | Up to 6 months
  PROPr gives health utility score integrating 7 domains (physical function, depression, fatigue, cognitive function, role satisfaction, sleep, and pain) using the PROMIS-29
  Scoring: Total scores range from 6 to 24, derived from 6 items scored on a 1-to-4 scale. Lower scores denote lower functional levels.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie P Scheunemann, MD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available from the PI upon request with a Data Use Agreement
Supporting Information: Study Protocol, ICF
Time Frame: Per any negotiated Data Use Agreement
Access Criteria: Negotiated Data Use Agreement

REFERENCES:
- [Background] LaMantia MA, Scheunemann LP, Viera AJ, Busby-Whitehead J, Hanson LC. Interventions to improve transitional care between nursing homes and hospitals: a systematic review. J Am Geriatr Soc. 2010 Apr;58(4):777-82. doi: 10.1111/j.1532-5415.2010.02776.x. PMID 20398162
- [Background] Polgar P, Taylor L. Alterations in prostaglandin synthesis during senescence of human lung fibroblasts. Mech Ageing Dev. 1980 Apr;12(4):305-10. doi: 10.1016/0047-6374(80)90063-9. PMID 6993800
- [Background] Bailey CL. The treatment of malaria. N Engl J Med. 1997 Mar 6;336(10):733; author reply 733-4. doi: 10.1056/NEJM199703063361017. No abstract available. PMID 9045053
- [Background] Scheunemann LP, Motter E, Kim SP, et al. Conceptualizing Transitional Care After Critical Illness Using Stakeholder Perspectives: A Qualitative Content Analysis. Under review. Published online 2023.
- [Background] Moale AC, Motter EM, Eisenhauer P, Gandhi N, Kim SP, Girard TD, Reynolds CF 3rd, Leland NE, Chang JC, Scheunemann LP. Integrating Perspectives on Family Caregiving After Critical Illness: A Qualitative Content Analysis. Am J Crit Care. 2024 May 1;33(3):180-189. doi: 10.4037/ajcc2024309. PMID 38688852
- [Background] Lewis A, Scheunemann LP, Roberts ET. Who, what, and where matter: Social determinants of health and functional outcomes in critical illness survivors. AcademyHealth Research Conference. Published online June 2022.
- [Background] Scheunemann LP, Leland NE, Perera S, Skidmore ER, Reynolds CF, Pandharipande PP, Jackson JC, Ely EW, Girard TD. Sex Disparities and Functional Outcomes after a Critical Illness. Am J Respir Crit Care Med. 2020 Apr 1;201(7):869-872. doi: 10.1164/rccm.201902-0328LE. No abstract available. PMID 31751152
- [Background] Scheunemann LP, Girard TD, Leland NE. Epidemiological Conceptual Models and Health Justice for Critically Ill Older Adults. Crit Care Med. 2021 Feb 1;49(2):375-379. doi: 10.1097/CCM.0000000000004793. No abstract available. PMID 33438978
- [Background] Naylor MD, Sochalski JA. Scaling up: bringing the transitional care model into the mainstream. Issue Brief (Commonw Fund). 2010 Nov;103:1-12. PMID 21053533
- [Background] Hirschman KB, Shaid E, McCauley K, Pauly MV, Naylor MD. Continuity of Care: The Transitional Care Model. Online J Issues Nurs. 2015 Sep 30;20(3):1. PMID 26882510
- [Background] Naylor MD, Brooten DA, Campbell RL, Maislin G, McCauley KM, Schwartz JS. Transitional care of older adults hospitalized with heart failure: a randomized, controlled trial. J Am Geriatr Soc. 2004 May;52(5):675-84. doi: 10.1111/j.1532-5415.2004.52202.x. PMID 15086645
- [Background] Naylor MD, Hirschman KB, Toles MP, Jarrin OF, Shaid E, Pauly MV. Adaptations of the evidence-based Transitional Care Model in the U.S. Soc Sci Med. 2018 Sep;213:28-36. doi: 10.1016/j.socscimed.2018.07.023. Epub 2018 Jul 17. PMID 30055423
- [Background] Skidmore ER, Swafford M, Juengst SB, Terhorst L. Self-Awareness and Recovery of Independence With Strategy Training. Am J Occup Ther. 2018 Jan/Feb;72(1):7201345010p1-7201345010p5. doi: 10.5014/ajot.2018.023556. PMID 29280726
- [Background] Berker F, Sandalci C, Ucer O. [Rare complication observed during the course of diabetes mellitus]. Turk Tip Cemiy Mecm. 1969;35(8):483-8. No abstract available. Turkish. PMID 5368028
- [Background] Dynovskii GD. [Late aftereffects of cranio-cerebral injuries]. Vrach Delo. 1974 Jun;(6):108-10. No abstract available. Russian. PMID 4466065
- [Background] Sendlmeier WF. [Speech processing in pathologic hearing. On the status of research]. Folia Phoniatr (Basel). 1988;40(5):218-43. No abstract available. German. PMID 3072282
- [Background] Sherr CJ. G1 phase progression: cycling on cue. Cell. 1994 Nov 18;79(4):551-5. doi: 10.1016/0092-8674(94)90540-1. No abstract available. PMID 7954821
- [Background] Higgins RJ, Randall CJ. Pasteurella multocida meningoencephalitis in a pheasant (Phasionus colchicus). Vet Rec. 1981 Apr 18;108(16):360. doi: 10.1136/vr.108.16.360. No abstract available. PMID 7269185
- [Background] Dewitt B, Feeny D, Fischhoff B, Cella D, Hays RD, Hess R, Pilkonis PA, Revicki DA, Roberts MS, Tsevat J, Yu L, Hanmer J. Estimation of a Preference-Based Summary Score for the Patient-Reported Outcomes Measurement Information System: The PROMIS(R)-Preference (PROPr) Scoring System. Med Decis Making. 2018 Aug;38(6):683-698. doi: 10.1177/0272989X18776637. Epub 2018 Jun 26. PMID 29944456
- [Background] Hanmer J, Dewitt B, Yu L, Tsevat J, Roberts M, Revicki D, Pilkonis PA, Hess R, Hays RD, Fischhoff B, Feeny D, Condon D, Cella D. Cross-sectional validation of the PROMIS-Preference scoring system. PLoS One. 2018 Jul 31;13(7):e0201093. doi: 10.1371/journal.pone.0201093. eCollection 2018. PMID 30063733
- [Background] The Accountable Health Communities Health-Related Social Needs Screening Tool. Center for Medicare and Medicaid Services
- [Background] Wallston KA, Cawthon C, McNaughton CD, Rothman RL, Osborn CY, Kripalani S. Psychometric properties of the brief health literacy screen in clinical practice. J Gen Intern Med. 2014 Jan;29(1):119-26. doi: 10.1007/s11606-013-2568-0. Epub 2013 Aug 6. PMID 23918160